CLINICAL TRIAL: NCT07083960
Title: An Open-Label, Phase 1b, Multiple Ascending Dose Study of OM336 in Participants With Active Autoimmune Cytopenias
Brief Title: OM336 in Autoimmune Cytopenias
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ouro Medicines (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OM336-AIC-1001
Record Dates: First submitted 2025-07-09; First posted 2025-07-24 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: AIHA - Warm Autoimmune Hemolytic Anemia; AIHA - Cold Autoimmune Hemolytic Anemia; ITP - Immune Thrombocytopenia
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune; Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OM336 Dose Escalation (Experimental): Participants will receive OM336 via subcutaneous injection in ascending dose cohorts
  Interventions: Drug: OM336

INTERVENTIONS:
Drug: OM336 — OM336 is an engineered bispecific antibody directed against BCMA and CD3

SUMMARY:
An early-phase clinical trial evaluating the safety, tolerability, and pharmacokinetics of subcutaneously dosed OM336 in adult participants with autoimmune cytopenias.

DETAILED DESCRIPTION:
An open-label, multicenter, ascending dose study, evaluating safety, tolerability, and PK/ADA of OM336 in autoimmune cytopenias.

ELIGIBILITY:
Key Inclusion Criteria:

* Active autoimmune cytopenia
* Relapsed/refractory after ≥1 prior treatment
* Body weight ≥ 55 kg
* Willing to comply with and study requirements and procedures

Key Exclusion Criteria:

* Previous treatment with a BCMA-targeted therapy
* Clinically significant infection within 3 months of screening
* Major surgery or splenectomy within 3 months of screening or planned during the study
* Pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 12 weeks
  Incidence and severity of treatment emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Safety and Tolerability | 52 weeks
  Incidence and severity of treatment-emergent adverse events (TEAEs)
To assess the pharmacokinetics (PK) of OM336 | 12 weeks
  Serum concentrations of OM336
Detection of anti-drug antibodies | 12 weeks
  Detection of anti-drug antibodies

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - The Canberra Hospital, Canberra, Australian Capital Territory
  - Liverpool Hospital, Sydney, New South Wales
  - Icon Cancer Center South Brisbane, Brisbane, Queensland

IPD SHARING:
Plan to Share IPD: No